CLINICAL TRIAL: NCT07164456
Title: Together Stronger: A Family-centered Lifestyle Intervention for Black Prostate Cancer Survivors and Their Caregivers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-0868; NCI-2025-06570 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-09-04; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Family Centered; Black Ethnicity; Prostate Cancer Survivors
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Family-centered intervention (Experimental): Includes a nutrition education session, a PA education session, and 12 health-coaching calls, all conducted via Zoom or phone.
  Interventions: Other: Education sessions; Other: Questionnaire
- survivor-only intervention (Experimental): Includes a nutrition education session, a PA education session, and 12 health-coaching calls, all conducted via Zoom or phone.
  Interventions: Other: Education sessions; Other: Questionnaire
- Health education control (Experimental): Will focus on enhancing participants' intrinsic motivation and problem-solving skills related to improving diet quality and engaging in PA. A total of 12 sessions will be provided, with approximately 2 sessions per month
  Interventions: Other: Education sessions; Other: Questionnaire

INTERVENTIONS:
Other: Education sessions — Remote and In person sessions
Other: Questionnaire — Questionnaires given a 3,6,12 mouth follow ups

SUMMARY:
To establish the efficacy of the family-centered intervention in improving healthy lifestyle behaviors (MVPA and overall diet quality), as well as physical functioning, QoL, and family health climate, compared to survivor-only and control groups.

DETAILED DESCRIPTION:
Primary Objectives

• Determine the extent to which MVPA and overall diet quality have improved in Black PCa survivors and their caregivers in the family-centered intervention group, compared to those in the survivor-only and control groups at post-intervention.

Secondary Objectives

* Determine the extent to which, compared to those in the survivor-only and control groups, both survivors and caregivers in the family-centered group maintain the MVPA and high diet quality at the 6-month follow-up, and experience improved 6MWT, QoL, and family health climate at both post-intervention and 6-month follow-up.
* Identify mediators and moderators of the family-centered intervention.

ELIGIBILITY:
Eligibility Criteria

Survivors are eligible if they

* Are adults (≥18 years old)
* Self-identify as Black or African American;
* Were diagnosed with stage 0-III PCa; completed PCa treatment; (5) are able to be physically active, as determined by responses to the Physical Activity Readiness Questionnaire (PAR-Q); and
* Have a family caregiver willing to participate together. Individuals under active surveillance for PCa will be included.

Caregivers are eligible if they:

* Are adults (≥18 years old)
* Are able to be physically active, as determined by responses to the

Exclusion Criteria

Survivors are excluded if they:

* Have a prior history of other cancer or have metastatic cancer.
* Have planned concomitant immunotherapy, hormonal therapy, chemotherapy, or radiation therapy during the study period.
* Meet physical activity recommendations (i.e., 150 min of moderate intensity physical activity per week); and (4) are currently participating in a lifestyle or weight management program.

Caregivers are excluded if they:

* Have serious medical conditions (e.g., cancer, congestive heart failure, stroke, and dementia)
* Are currently participating in a lifestyle or weight management program.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — males
Enrollment: 648 (Estimated)
Dates: Start 2026-02-14 (Estimated); Primary Completion 2031-06-30 (Estimated); Study Completion 2033-06-30 (Estimated)

PRIMARY OUTCOMES:
Physical Activity Readiness Questionnaire | Through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dalnim Cho, MD, Principal Investigator — MD Andersson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org